CLINICAL TRIAL: NCT03912870
Title: Interest of Flow Cytometry in Infectious Point of Care: Feasibility Study
Brief Title: Value of Flow Cytometry in Infectious Point of Care: Feasibility Study
Status: Completed | Type: Observational
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-62
Record Dates: First submitted 2019-04-10; First posted 2019-04-11 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: A Potential Infectious Respiratory Clinical Syndrome; Potential Clinical Urinary Infectious Syndrome; A Potential Clinical Abdominal Infection Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Value of Flow Cytometry in Infectious Point of Care — To validate the diagnostic orientation properties of two new biomarkers (CD64, CD169) for patients with infectious syndromes arriving in emergency departments. This prospective observational study will focus on the quantification of these biomarkers on a hematology tube background (Pr Morange laboratory) without modifying the usual diagnostic and therapeutic procedures. The results of these assays will be compared with the diagnoses made at the end of treatment in order to determine their sensitivity and specificity.
  This study is the preliminary study, necessary to determine the detection characteristics of these biomarkers.

SUMMARY:
The purpose of this project is to validate the diagnostic orientation properties of two new biomarkers (CD64, CD169) for patients with infectious syndromes arriving in emergency departments. This prospective observational study will focus on the quantification of these biomarkers on a hematology tube background (Pr Morange laboratory) without modifying the usual diagnostic and therapeutic procedures. The results of these assays will be compared with the diagnoses made at the end of treatment in order to determine their sensitivity and specificity.

This study is the preliminary study, necessary to determine the detection characteristics of these biomarkers.

DETAILED DESCRIPTION:
The detection and characterization of infectious events is a major challenge for emergency medicine. Thus the possibility of quickly attributing an infectious origin to a febrile and/or inflammatory syndrome makes it possible to treat and refer the patient quickly. In addition, the ability to distinguish bacterial etiology from viral etiology provides a valuable additional indication for the clinician. This of the upmost importance for fragile populations such as elderly patients and in epidemic conditions such as influenza. A new rapid diagnostic guidance solution is proposed by the Beckman Coulter Laboratory with the simultaneous assay of two biomarkers, one allowing the detection of a viral infectious process (CD169), the other of a bacterial infectious process (CD64). The combination of these two biomarkers, measured in 12 minutes by a new generation assay and flow cytometer, represents an opportunity for emergency services.

To date, there is no study on the validation of this diagnostic orientation method. We propose to carry out a prospective, observational, non-interventional feasibility study to compare the results of these measurements with the usual diagnostic criteria combining the clinical signs, infectious testing, and biological data.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years of age presenting to the Timone 2 Emergency Department with the association:

  * A fever> 38 ° C or hypothermia <36.5 ° C.
  * A potential clinical infectious syndrome is respiratory (cough, sputum, dyspnea), or urinary (potential urinary tract infection), or abdominal (potentially infectious diarrhea, potentially infectious pain syndrome) or neurological (meningitis potential) or cutaneous (erysipelas).

Exclusion Criteria:

* Patients with clinical criteria that may increase other non-specific biomarkers and therefore not allow for subsequent comparison:

  * Trauma
  * Known inflammatory and autoimmune disease
  * Infectious chronic viral, fungal or bacterial disease
  * Antibiotic or anti viral treatment prior to admission
  * Immunosuppressive treatment
  * neoplasia
  * Extended burn
  * Recent surgery (<1 month)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient over 18 years of age presenting to the Timone 2 Emergency Department with the association
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2018-12-10 (Actual); Primary Completion 2020-06-05 (Actual); Study Completion 2023-05-11 (Actual)

PRIMARY OUTCOMES:
Variables specifically measured for this study will be the flow cytometry assay of the two biomarkers (CD64, CD169) | 96 hours
  to validate the diagnostic orientation properties of two new biomarkers (CD64, CD169) for patients with infectious syndromes arriving in emergency departments. This prospective observational study will focus on the quantification of these biomarkers on a hematology tube background (Pr Morange laboratory) without modifying the usual diagnostic and therapeutic procedures

CONTACTS AND LOCATIONS:
Overall Officials: Pierre MICHELET, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France